CLINICAL TRIAL: NCT03923127
Title: PJ-013483 FLAGSHIP Transitional Care Study 3
Brief Title: Transitional Care Study 3
Acronym: TRICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ICBE-2-27377
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Surgery--Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elan and HealthDot (Experimental): Patients with elective surgery will wear two devices (HealthDot and Elan) after surgery in hospital and after discharge at home for up to 2 weeks (HealthDot) or 3 weeks (Elan).
  Interventions: Other: Elan and HealthDot

INTERVENTIONS:
Other: Elan and HealthDot — Patients with elective surgery will wear two devices (HealthDot and Elan) after surgery in hospital and after discharge at home for up to 2 weeks (HealthDot) or 3 weeks (Elan).

SUMMARY:
In this study patients with elective surgery will wear two devices (HealthDot and Elan) after surgery in hospital and after discharge at home for up to 2 weeks (HealthDot) or 3 weeks (Elan). The HealthDot will measure heart rate, posture, activity and respiratory rate which are stored on the device as well as sent to Philips. The Elan device will measure PPG and accelerometer data which is transferred to Philips. The data collected will be used for algorithm development. Data will be analysed retrospectively and compared to readmission and adverse events to see if the events could have been predicted due to the collected data by the devices. No clinical decisions will be based on the measurements done during the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Willing and able to sign informed consent form
* Willingness to abstain from visiting a sauna during the study period
* Willingness to dry area where the HealthDot is applied in a dipping fashion after washing
* Willingness to abstain from flying during the study period of time
* Elective surgery
* General anesthesia required for surgery

Exclusion Criteria:

* General inmates of psychiatric wards, prisons, or other state institutions
* Investigator or any other team member involved directly or indirectly in the conduct of the clinical study
* Any skin condition, for example prior rash, discoloration, scars or open wounds at the area of investigation of both devices
* Pregnant, or breastfeeding
* Known to be allergic for the tissue adhesive used in the HealthDot.
* Use of topical that is known to influence the skin at the test area (such as medical and non-medical creams or lotions)
* Patient with active implantables such as Implantable Cardioverter Defibrilator (ICD) and pacemaker
* Unable to understand instructions
* Expected participation less than 2 weeks
* Left lower rib (place where HealthDot will be applied) is involved in the area of surgery, area of disinfection or area where bandages are needed.
* Area on arm where the Elan device is applied is involved in the surgical procedure.
* Patients with antibiotic resitant infections (e.g. MRSA).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity | 3 weeks
  Evaluate the sensitivity and specificity for the prediction of deterioration after surgery using the data from both devices.

SECONDARY OUTCOMES:
Accuracy HealthDot | 2 weeks
  Evaluate if the calculated heart rate and respiratory rate data collected by HealthDot are accurate compared to a gold standard as used in the hospital
Comfort of wearing measured by questionnaire | at week 2
  Comfort of wearing the HealthDot will be assessed by VAS scale 1-10 while 1 beeing very comfortable, and 10 very uncomfortable
Accuracy Elan | 3 weeks
  Evaluate if the calculated heart rate and respiratory rate data collected by Elan are accurate compared to a gold standard as used in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Eveline Mestrom, Principal Investigator — Catharina Hospital, Eindhoven, The Netherlands
Locations (1):
- Catharina Hospital, Eindhoven, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van der Stam JA, Mestrom EHJ, Scheerhoorn J, Jacobs FENB, Nienhuijs S, Boer AK, van Riel NAW, de Morree HM, Bonomi AG, Scharnhorst V, Bouwman RA. The Accuracy of Wrist-Worn Photoplethysmogram-Measured Heart and Respiratory Rates in Abdominal Surgery Patients: Observational Prospective Clinical Validation Study. JMIR Perioper Med. 2023 Feb 20;6:e40474. doi: 10.2196/40474. PMID 36804173